CLINICAL TRIAL: NCT05581251
Title: The Relationship Between Food and Cooking Skills, and Eating Behaviors in People With Overweight or Obesity
Brief Title: Food and Cooking Skills, and Eating Behaviors in People With Overweight or Obesity
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sedat Arslan, Assistant Professor, Hacettepe University
Other Study IDs: STUDY020265
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Overweight
Keywords: food skills; cooking skills; eating behavior
MeSH Terms: conditions — Obesity; Overweight; Feeding Behavior | interventions — Food

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Food and cooking skills — The researchers collected the study data using the face-to-face interview method through a questionnaire including the Descriptive Information Form, Cooking Skills and Food Skills Scale, and Three-Factor Eating Questionnaire-R21.

SUMMARY:
In the present study, the authors aimed to determine food skills and cooking skills, and eating behaviors, and to evaluate the relationship between food skills and cooking skills, and eating behaviors in people with overweight or obesity.

Methods: This cross-sectional study was conducted with 185 people with overweight or obesity. The researchers collected the study data using the face-to-face interview method through a questionnaire including the Descriptive Information Form, Cooking Skills and Food Skills Scale, and Three-Factor Eating Questionnaire-R21. Numbers, percentages, arithmetic mean, standard deviation, Student's t-test, Pearson Chi-Square test, and multiple linear regression analysis were used in the analysis of the data.

DETAILED DESCRIPTION:
Food skills and cooking skills, considered a basic activity of daily living, have become an increasingly important issue, especially in Western countries in parallel with the change in food consumption patterns such as consuming Away-From-Home-Food and processed food. Food skills which include concepts such as menu planning for meals, purchasing, preparing and cooking foods, budgeting, food safety, and healthy nutrition using the resources at hand are defined as "the ability to produce balanced and delicious meals suitable for the age and needs of individuals". Cooking skills not only refer to a series of mechanical or physical skills such as chopping, mixing, and heating used in food preparation but also include conceptual and perceptual skills related to changes in food after the cooking process. The increase in obesity on a global scale and the significant decline in diet quality draw attention to the issue of increasing people's interest in home cooking and methods of preparing food to be eaten at home as a potential strategy for preventing obesity. Thus, it is stated that food preparation knowledge, skills, and behaviors can affect dietary intake and body weight.

This study cross-sectional was conducted in the Nutrition and Diet Clinic of Bandirma Training and Research Hospital in Bandirma district of Balikesir province, located on the coast of the Marmara Sea, in the west of Turkey. The minimum sample size was calculated as 107 using the G*Power 3.1.9.7 program (power:95%, α=0.05, effect size d=0.15). However, considering the possibility of losses during the study, we decided to include 30% (n = 139) more people.

Of the individuals who presented to the diet outpatient clinic between January 2022 and July 2022, those who agreed to participate in the study (n=308), were in the age group of 19-64 years (n=212) and had a Body Mass Index (BMI) of 25.00 kg/m2 were included in the study. Written informed consent was obtained from the participants. Of these individuals, those with a diagnosis of psychiatric disease (n=8), those who cannot feed orally and/or have difficulty in chewing and swallowing (n=4), and those who had physical health problems that would prevent the researchers from assessing their food preparation and cooking skills or from making their anthropometric measurements (n=13) and those who were pregnant or lactating (n=2) were excluded, and data about 185 individuals were evaluated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Obesity
* who were in the age group of 19-64 years

Exclusion Criteria:

* Clinical diagnosis of psychiatric disease
* Who cannot feed orally and/or have difficulty in chewing and swallowing
* Who had physical health problems that would prevent the researchers from assessing their food preparation and cooking skills or from making their anthropometric measurements
* Who were pregnant or lactating

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study cross-sectional was conducted in the Nutrition and Diet Clinic of Bandirma Training and Research Hospital in Bandirma district of Balikesir province, located on the coast of the Marmara Sea, in the west of Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
In people with overweight or obesity, cognitive restraint and emotional eating behaviors improve as their food preparation and cooking skills improve. | 6 months
  The researchers collected the study data using the face-to-face interview method through a questionnaire including the Descriptive Information Form, Cooking Skills and Food Skills Scale, and Three-Factor Eating Questionnaire-R21.
  In order to measure the BMI values of the individuals who presented to the Nutrition and Diet Clinic, the researchers who were experts in the field of nutrition and dietetics used a 100-gram precision SECA brand portable digital scale. During the measurements, the individuals wore light clothes and took off their shoes. Their height was measured in centimeters (cm) using a portable height-measuring rod with a 1-mm precision. The height-measuring rod can measure heights between 14 and 200 cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeni mh. Bandirma Onyedi Eylul University Faculty of Health Science Bandirma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No